CLINICAL TRIAL: NCT01835912
Title: Chronic vs. Acute Ingestion of Sodium Citrate: a Randomised Placebo Controlled Cross-over Trial for Swimming a 200 Metres in Well-trained Swimmers Age 13-17
Brief Title: Chronic Versus Acute Dosing of Sodium Citrate for Swimming 200m
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Colin Russell, M.Sc. Researcher Brock University, Brock University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 12-009
Record Dates: First submitted 2013-04-10; First posted 2013-04-19 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Alkalosis
Keywords: performance; speed; exertion
MeSH Terms: conditions — Alkalosis | interventions — Sodium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Flavoured water placebo for acute dosing (Placebo Comparator): 500 milliliters flavoured water (placebo for the acute dosing intervention of sodium citrate)
  Interventions: Other: Sodium Citrate Dihydrate
- Sodium Citrate Dihydrate Acute (Experimental): dose: 0.5 g/kg of body mass dissolved in 500 milliliters of flavoured water
  Interventions: Other: Sodium Citrate Dihydrate
- Flavoured water placebo chronic dosing (Placebo Comparator): 500 milliliters flavoured water (placebo for the chronic dosing intervention of sodium citrate)
  Interventions: Other: Sodium Citrate Dihydrate
- Sodium Citrate Dihydrate Chronic (Experimental): 3 days of 0.1g/kg of body mass of sodium citrate and 4th day at 0.3 g/kg of body mass of sodium citrate in 500 milliliters of flavoured water
  Interventions: Other: Sodium Citrate Dihydrate

INTERVENTIONS:
Other: Sodium Citrate Dihydrate — Dose sodium citrate dihydrate through 2 dosing protocols (Acute and Chronic)
  Other Names: CAS: 6132-04-3

SUMMARY:
Ingestion of sodium citrate (Na-Cit), an alkalizing agent, increases extracellular pH via liver oxidation by decreasing [H+] and increasing bicarbonate concentration (HCO3-). Studies have confirmed that increasing extracellular pH promotes the efflux of La- and H+ from active muscles. This is due to an increase in activity of the pH sensitive monocarboxylate transporter as the gradient of intracellular versus extracellular H+ increases. Therefore, artificially inducing alkalosis prior to anaerobic exercise may reduce intracellular acidosis and increase the time to fatigue - defined as a decrease in force production with an increased perception of effort. The investigators will test the null hypothesis that sodium citrate ingestion (chronic and acute) will not have an effect on exercise performance compared to placebo.

DETAILED DESCRIPTION:
Anaerobic glycolysis quickly provides adenosine triphosphate (ATP) for muscular contraction during high intensity, short duration exercise. The fast rate of glycolysis during anaerobic exercise results in pyruvate formation exceeding pyruvate oxidation resulting in a build up of lactic acid. Lactic acid dissociates quickly to lactate (La-) and hydrogen ion (H+) which causes a decrease in muscle and blood pH. The increase in H+ causes impaired release of calcium from the sarcoplasmic reticulum and calcium ion binding which inhibits the coupling of actin and myosin.

Ingestion of sodium citrate (Na-Cit), an alkalizing agent, increases extracellular pH via liver oxidation by decreasing [H+] and increasing bicarbonate concentration (HCO3-). Studies have confirmed that increasing extracellular pH promotes the efflux of La- and H+ from active muscles. This is due to an increase in activity of the pH sensitive monocarboxylate transporter as the gradient of intracellular versus extracellular H+ increases. Therefore, artificially inducing alkalosis prior to anaerobic exercise may reduce intracellular acidosis and increase the time to fatigue - defined as a decrease in force production with an increased perception of effort. Furthermore, Cit- enters the cell through the Plasma Membrane Citrate Transporter and in the cell Cit- is involved in a number of processes: i) intermediary in the Krebs Cycle, ii) transports acetyl-Co-enzyme A (CoA)from the mitochondria to the cytosol for fatty-acid synthesis, iii) negative allosteric effector of phosphofructokinase, iv) anionic effect on membrane potential can cause a reduction in the contraction threshold.

Researchers have studied sodium bicarbonate and Na-Cit as potential alkalizing agents. Na-Cit has been studied in few sports over a broad array of doses, times, and distances with inconclusive results. McNaughton et al. researched the optimal doses and durations for Na-Cit to be potentially beneficial to performance. They concluded that 0.3-0.5g/kg, 90-120 minutes prior to maximal effort are the optimal conditions for potential ergogenic effect. The only reported side effect was gastrointestinal (GI) discomfort in a 3 of the 8 subjects. However, it seems Na-Cit is handled better than the more commonly employed sodium bicarbonate.

The investigators will test the null hypothesis that sodium citrate ingestion (chronic and acute) will not have an effect on exercise performance compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17
* Male
* Regional, provincial and national level swimmers

Exclusion Criteria:

* Females
* Level of swimming below regional level standards
* Caffeine before trials
* Chronic health concerns
* Health problems before or during the course of the trial

Ages: 13 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nota Klentrou, PhD, Study Director — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

REFERENCES:
- [Derived] Russell C, Papadopoulos E, Mezil Y, Wells GD, Plyley MJ, Greenway M, Klentrou P. Acute versus chronic supplementation of sodium citrate on 200 m performance in adolescent swimmers. J Int Soc Sports Nutr. 2014 Jun 12;11:26. doi: 10.1186/1550-2783-11-26. eCollection 2014. PMID 24944546

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Sodium Citrate Dihydrate: Dose sodium citrate dihydrate through 2 dosing protocols (Acute and Chronic) and their corresponding placebos.
  4 arms: Acute, Acute Placebo, Chronic, Chronic Placebo
  Acute: 0.5 g/kg of body mass of sodium citrate in 500 millilitres of flavoured water
  Acute Placebo: 500 milliliters of flavoured water
  Chronic: 3 days of 0.1 g/kg of body mass of sodium citrate and 4th day at 0.3 g/kg of body mass of sodium citrate in 500 millilitres of flavoured water
  Chronic Placebo: 3 days of 500 millilitres of flavoured water and 4th day 500 millilitres of flavoured water
Period: Overall Study
Arm/Group | All Study Participants
Started | 10
Acute | 10
Acute Placebo | 10
Chronic | 10
Chronic Placebo | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Acute: dose: 0.5 g/kg of body mass dissolved in 500 milliliters of flavoured water
  Sodium Citrate Dihydrate: Dose sodium citrate dihydrate through 2 dosing protocols (Acute and Chronic)
  Acute Placebo: 500 milliliters flavoured water (placebo for the acute dosing intervention of sodium citrate)
  Chronic: 3 days of 0.1g/kg of body mass of sodium citrate and 4th day at 0.3 g/kg of body mass of sodium citrate in 500 milliliters of flavoured water
  Sodium Citrate Dihydrate: Dose sodium citrate dihydrate through 2 dosing protocols (Acute and Chronic)
  Chronic Placebo: 3 days of 500 milliliters flavoured water and the 4th day 500 milliliters flavoured water (placebo for the chronic dosing intervention of sodium citrate)
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  males | 10
Region of Enrollment [Number; unit: participants]
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Time
Description: time to complete 200 metre swimming performances in seconds
  Participants chose type of swim stroke to swim a maximal effort 200 metre performance
Time Frame: once each 200m performance
Measure: Mean (Standard Error); unit: seconds
Groups:
- Flavoured Water Placebo for Chronic Dosing: 500 milliliters flavoured water (placebo for the chronic dosing intervention of sodium citrate)
Arm/Group | Flavoured Water Placebo for Acute Dosing | Sodium Citrate Dihydrate Acute | Flavoured Water Placebo for Chronic Dosing | Sodium Citrate Dihydrate Chronic
Number analyzed (Participants) | 10 | 10 | 10 | 10
seconds | 144.2 (4.7) | 145.3 (5.3) | 145.3 (5.4) | 144.8 (5.3)

2. Secondary Outcome: Lactate
Description: lactate measured at 3min post trial
Time Frame: 3 min post performance
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Flavoured Water Placebo for Acute Dosing | Sodium Citrate Dihydrate Acute | Flavoured Water Placebo for Chronic Dosing | Sodium Citrate Dihydrate Chronic
Number analyzed (Participants) | 10 | 10 | 10 | 10
mmol/L | 8.8 (0.7) | 10.4 (1.3) | 9.5 (1.2) | 10.8 (1)

3. Other Pre Specified Outcome: Rate of Perceived Exertion
Description: Rate of perceived exertion (RPE) was recorded after each 200 metre swimming performance
  RPE scale is from 6-20. Minimum = 6 (level of exertion equal to lying down) and Maximum = 20 (maximal perceived exertion)
  Numbers reported are the average of the RPE recorded for all 10 participants.
Time Frame: Rate of Perceived Exertion after each 200m swimming performance
Measure: Mean (Standard Error); unit: units on a scale (6-20)
Arm/Group | Flavoured Water Placebo for Acute Dosing | Sodium Citrate Dihydrate Acute | Flavoured Water Placebo for Chronic Dosing | Sodium Citrate Dihydrate Chronic
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale (6-20) | 16.4 (0.6) | 16.1 (0.6) | 16.6 (0.3) | 17.1 (0.6)

ADVERSE EVENTS:
Arm/Group | Flavoured Water Placebo for Acute Dosing | Sodium Citrate Dihydrate Acute | Flavoured Water Placebo for Chronic Dosing | Sodium Citrate Dihydrate Chronic
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No